CLINICAL TRIAL: NCT05753657
Title: A Pilot Study of Monitoring Insulin Levels and Treating Hyperinsulinemia and Hyperglycemia With Pioglitazone in Patients Treated With Alpelisib for Metastatic Breast Cancer.
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Ayelet Shai MD, Head of breast cancer unit, Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0494-22-RMB
Record Dates: First submitted 2022-12-26; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Breast Cancer; Hyperinsulinism; Hyperglycemia Drug Induced
MeSH Terms: conditions — Breast Neoplasms; Hyperinsulinism | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): treating hyperinsulinemia and hyperglycemia with pioglitazone in patients treated with Alpelisib for metastatic breast cancer
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — hyperinsulinemia and hyperglycemia

SUMMARY:
The goal of this study is to test whether monitoring insulin levels and using pioglitazone to treat hyperglycemia and hyperinsulinemia in patients treated with Alpelisib for metastatic breast cancer is feasible and safe, and to assess the rates of glycemic control, dose reductions and treatment discontinuation and the progression free survival of patients treated with this regimen.

DETAILED DESCRIPTION:
1. To assess the feasibility and safety of monitoring insulin levels alongside glucose levels and of directing antidiabetic treatment according to insulin and fasting glucose levels in patients treated with Alpelisib for metastatic breast cancer.
2. To assess the feasibility and safety of treatment with pioglitazone in these patients.
3. To assess the rate of severe (grade 3-4) hyperglycemia in patients treated according to this protocol.
4. To assess the rates of dose reductions and treatment discontinuation due to hyperglycemia in patients treated according to this protocol.
5. To assess the median progression free survival of patients treated according to this protocol

ELIGIBILITY:
Inclusion Criteria:

* Patients with ER positive HER2 negative metastatic breast cancer, harboring an activating PIK3CA mutation, scheduled to start treatment with Alpelisib and fulvestrant.
* Ages 18 - 85
* ECOG performance status 0, 1 or 2
* Ability to understand and willingness to sign a written informed consent.

Exclusion Criteria:

* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of Alpelisib
* Uncontrolled diabetes mellitus, defined as HbA1c above 8%
* Diabetes mellitus controlled by insulin
* Uncontrolled intercurrent illness including, but not limited to: active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnancy
* Known allergy to pioglitazone

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of severe (grade 3 and 4) hyperglycemia in patients enrolled in the study and in patients treated per protocol | through study completion, an average of 1 year
Rate of all grade hyperglycemia in patients enrolled in the study and in patients treated per protocol | through study completion, an average of 1 year
Progression free survival in patients enrolled in the study and in patients treated per protocol | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ayelet Shai, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No